CLINICAL TRIAL: NCT03836209
Title: Randomized Trial of Gilteritinib vs Midostaurin in FLT3 Mutated Acute Myeloid Leukemia (AML)
Brief Title: Gilteritinib vs Midostaurin in FLT3 Mutated Acute Myeloid Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: PrECOG, LLC. (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PrE0905
Record Dates: First submitted 2019-02-07; First posted 2019-02-11 (Actual); Results first posted 2025-02-28 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Acute Myeloid Leukemia
Keywords: Gilteritinib; Midostaurin; Daunorubicin; Cytarabine; FLT3; FLT3 Mutation; FLT3 Internal Tandem Duplication (ITD); FLT3 ITD; FLT3 Tyrosine Kinase Domain (TKD); FLT3 TKD
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — gilteritinib; midostaurin; Daunorubicin; Cytarabine

STUDY DESIGN:
Intervention Model Description: Open-Label, Randomized trial of Daunorubicin/Cytarabine and High Dose Cytarabine + Gilteritinib vs Midostaurin for Induction and Consolidation. FLT3 mutated patients will be stratified based on TKD vs ITD. Patients who are FLT3 ITD will be further stratified by Signal Ratio (high vs. low of FLT3 Wild Type) and Nucleophosmin 1-Mutated (NPM1) [positive vs negative].
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Experimental): Induction: Daunorubicin, cytarabine and gilteritinib. Depending on response, second cycle of Induction may be given.
  Consolidation: High-dose cytarabine and gilteritinib.
  Interventions: Drug: Gilteritinib; Drug: Daunorubicin; Drug: Cytarabine
- Arm B (Active Comparator): Induction: Daunorubicin, cytarabine and midostaurin. Depending on response, second cycle of Induction may be given.
  Consolidation: High-dose cytarabine and midostaurin.
  Interventions: Drug: Midostaurin; Drug: Daunorubicin; Drug: Cytarabine

INTERVENTIONS:
Drug: Gilteritinib — Induction: 120 mg orally daily x 14 days starting on day 8
  Consolidation: 120 mg orally daily x 14 days starting on day 8 of each cycle (up to 4 cycles)
  Other Names: ASP2215
  Arms: Arm A
Drug: Midostaurin — Induction: 50 mg orally twice daily x 14 days beginning on day 8
  Consolidation: 50 mg orally twice daily x 14 days beginning on day 8 of each cycle (up to 4 cycles)
  Other Names: RYDAPT
  Arms: Arm B
Drug: Daunorubicin — First Induction: Daunorubicin 90 mg/m²/day IV Days 1,2,3
  Second Induction, if needed: Daunorubicin 45 mg/m²/day IV Days 1,2,3
  Other Names: Daunorubicin hydrochloride; Daunomycin; Rubidomycin; Cerubidine
Drug: Cytarabine — Induction: Cytarabine 100 mg/m²/day continuous infusion x 7 days starting Day 1
  Second Induction, if needed: Cytarabine 100 mg/m²/day continuous infusion x 7 days starting Day 1
  Consolidation: Cytarabine 3 g/m² (recommend 1.5 g/m² for age ≥ 55 or patients with decreased creatinine clearance) every 12 hours IV Days 1,3,5 or Days 1-3 for 6 doses for up to 4 cycles
  Other Names: Cytosar-U; Ara-C; Arabinosyl; Cytosine Arabinoside

SUMMARY:
Eligible untreated patients with FLT3 acute myeloid leukemia (AML) between the ages of 18 and 70 will be randomized to receive gilteritinib or midostaurin during induction and consolidation. Patients will also receive standard chemotherapy of daunorubicin and cytarabine during induction and high-dose cytarabine during consolidation.

Gilteritinib, is an oral drug that works by stopping the leukemia cells from making the FLT3 protein. This may help stop the leukemia cells from growing faster and thus may help make chemotherapy more effective. Gilteritinib has been approved by the Food and Drug Administration (FDA) for patients who have relapsed or refractory AML with a FLT3 mutation but is not approved by the FDA for newly diagnosed FLT3 AML, and its use in this setting is considered investigational.

Midostaurin is an oral drug that works by blocking several proteins on cancer cells, including FLT3 that can help leukemia cells grow. Blocking this pathway can cause death to the leukemic cells. Midostaurin is approved by the FDA for the treatment of FLT3 AML.

The purpose of this study is to compare the effectiveness of gilteritinib to midostaurin in patients receiving combination chemotherapy for FLT3 AML.

DETAILED DESCRIPTION:
Approximately one third of patients with AML have a particular change in their leukemia cells (called a mutation) in a gene called FLT3. The presence of a FLT3 mutation can be used to direct treatment options.

This is an open-label phase II study. Patients will receive standard chemotherapy of daunorubicin and cytarabine during Induction and high-dose cytarabine during Consolidation. Patients will be randomized to gilteritinib or midostaurin. After approximately 90 patient's complete treatment, a review of the effectiveness of gliteritinib compared to midostaurin will be done. If gilteritinib is not as effective as midostaurin, the study may be stopped.

Bone marrow aspirate and biopsy will be done on Day 21 after start of Induction and after Induction to assess response. Patients with a complete response may proceed to consolidation chemotherapy. Another bone marrow aspirate and biopsy will be done after the first cycle of consolidation is complete.

Mandatory prescreening bone marrow and/or blood samples are required for FLT3 testing. Any left-over samples will be requested for future research (optional).

Mandatory bone marrow samples for research are required after Induction and if patient receives Consolidation, after the first cycle of Consolidation.

ELIGIBILITY:
Registration Criteria:

* Any patient undergoing bone marrow biopsy with suspicion of or known diagnosis of acute myeloid leukemia (AML) will be asked to sign a Prescreening Consent to allow for centralized testing of bone marrow/peripheral blood samples.

Randomization Eligibility Criteria:

* Patient must have previously untreated FLT3 mutated Non M3 AML (FLT3-TKD or FLT3-ITD allowed).

  ° Standard of care induction 7+3 chemotherapy may start prior to randomization using same regimen and doses as defined in the protocol while awaiting prescreening test results.
* Patient must have had no prior systemic therapy for AML, except as noted below:

  * Hydroxyurea and emergent leukapheresis or preemptive treatment with retinoic acid prior to exclusion of Acute Promyelocytic Leukemia (APL) allowed.
  * Prior therapy for myelodysplastic syndrome (MDS) or myeloproliferative neoplasms (MPN) (e.g., thalidomide or lenalidomide, interferon, jakafi, cytokines, 5-azacytidine or decitabine, histone deacetylase inhibitors).
  * Initiation of standard of care 7+3 induction chemotherapy using same regimen and doses as defined in protocol while awaiting prescreening test results
* Patient may not have received hypomethylating agent within 21 days.
* Patient may not have M3 AML.
* Patient may not have AML with known Core Binding Factor -t(8;21), inv(16), t(16;16).
* Patient may not have known active Central Nervous System (CNS) leukemia.

  ° Prophylaxis with intrathecal chemotherapy is allowed prior to or during induction/consolidation.
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-3.
* Patient must be age ≥ 18 years to ≤ 70 years.
* Patient must be able to understand and willing to sign Institutional Review Board (IRB)-approved informed consent.
* Patient must be willing to provide mandatory bone marrow and blood samples for research.
* Patient must have adequate organ function as measured by the following criteria, obtained ≤ 48 hours prior to randomization except ECG and left ventricular ejection fraction (LVEF) which can be done ≤ 2 weeks prior to randomization:

  * Serum creatinine ≤ 1.5x institutional upper limit of normal (ULN), or if serum creatinine outside normal range, then glomerular filtration rate (GFR) >40 mL/min as measured by Cockcroft-Gault formula.
  * Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) ≤ 3x ULN, unless secondary to leukemia.
  * Serum total or direct bilirubin <2 mg/dL, unless due to Gilbert's, hemolysis or leukemic infiltration.
  * Fridericia-Corrected QT Interval (QTcF) interval ≤ 500 msec (using Friderica's correction).
  * Left Ventricular Ejection Fraction >45%.
* The patient may not be known to have hypokalemia and/or hypomagnesemia that does not respond to supplementation.
* A female patient is eligible to participate if she is not pregnant and at least one of the following conditions apply:

  * Not a woman of childbearing potential (WOCBP) OR
  * WOCBP who agrees to follow the contraceptive guidance throughout the treatment period and for at least 180 days after the final study drug administration.
* Female patient must agree not to breastfeed or donate ova starting at treatment and throughout the study period, and for at least 180 days after the final study drug administration.
* A male patient must agree not to donate sperm starting at treatment and throughout the study period, and for at least 120 days after the final study drug administration.
* A male patient with female partner(s) of child-bearing potential must agree to use contraception during the treatment period, and for at least 120 days after the final study drug administration.
* Male patient with a pregnant or breastfeeding partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy or time partner is breastfeeding throughout the treatment period, and for at least 120 days after the final study drug administration.
* Patient may not have another malignancy that could interfere with the evaluation of safety or efficacy of this combination.
* Patient may not have a history of Long QT Syndrome.
* Patient may not have evidence of uncontrolled angina, severe uncontrolled ventricular arrhythmias, electrocardiographic evidence of acute ischemia, or congestive heart failure (CHF) New York Heart Association (NYHA) Class 3 or 4. Patient may also not have a history of CHF NYHA Class 3 or 4 in the past, unless a prescreening echocardiogram (ECHO) or multigated acquisition scan (MUGA) performed within 2 weeks prior to study entry with results of left ventricular ejection fraction >45%.
* Patient may not have had major surgery or radiation therapy within 4 weeks of registration.
* Patient may not require treatment with concomitant drugs that are strong inducers of CYP3A and P-gp.
* Patient with a known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent are not eligible.
* Patient with known gastrointestinal (GI) disease or prior GI procedure that could interfere with the oral absorption or tolerance of gilteritinib or midostaurin including difficulty swallowing are not eligible.
* Patient with any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of the treatment according to the protocol are not eligible.
* Patient may not participate in any other therapeutic clinical trials, including those with other investigational agents not included in this trial during treatment on this study without prior approval from PrECOG.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2026-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Selena Luger, MD, Study Chair — University of Pennsylvania
Locations (44):
- United States (44):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - University of California, San Francisco-Fresno (University Oncology Associates), Clovis, California
  - UCLA, Los Angeles, California
  - Kaiser Permanente Oakland, Oakland, California
  - UC Irvine Health, Orange, California
  - Kaiser Permanente Roseville, Roseville, California
  - Kaiser Permanente Santa Clara, Santa Clara, California
  - Mayo Clinic- Jacksonville, FL, Jacksonville, Florida
  - Augusta University Medical Center, Augusta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - University of Kentucky Markey Cancer Center, Lexington, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - St. Joseph's Mercy Hospital, Ann Arbor, Michigan
  - Mayo Clinic- Rochester, MN, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Atlantic Health Systems/Morristown Medical Center, Morristown, New Jersey
  - Northwell Health, Lake Success, New York
  - Mount Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medicine New York Presbyterian Hospital, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - East Carolina University, Greenville, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - University of Oklahoma Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - LDS Hospital, Salt Lake City, Utah
  - MultiCare, Spokane, Washington
  - West Virginia University, Morgantown, West Virginia
  - University of Wisconsin Clinical Science Center, Madison, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin

IPD SHARING:
Plan to Share IPD: No
Data is proprietary.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All randomized, eligible, and treated patients.
  3 patients passed away/withdrew before induction. 1 patient determined to not have the diagnosis to meet the eligibility criteria and was removed from the study (181 consented).
Groups:
- Arm A: Induction: Daunorubicin, cytarabine and gilteritinib. Depending on response, second cycle of Induction may be given.
  Consolidation: High-dose cytarabine and gilteritinib.
  Gilteritinib: Induction: 120 mg orally daily x 14 days starting on day 8
  Consolidation: 120 mg orally daily x 14 days starting on day 8 of each cycle (up to 4 cycles)
  Daunorubicin: First Induction: Daunorubicin 90 mg/m²/day IV Days 1,2,3
  Second Induction, if needed: Daunorubicin 45 mg/m²/day IV Days 1,2,3
  Cytarabine: Induction: Cytarabine 100 mg/m²/day continuous infusion x 7 days starting Day 1
  Second Induction, if needed: Cytarabine 100 mg/m²/day continuous infusion x 7 days starting Day 1
  Consolidation: Cytarabine 3 g/m² (recommend 1.5 g/m² for age ≥ 55 or patients with decreased creatinine clearance) every 12 hours IV Days 1,3,5 or Days 1-3 for 6 doses for up to 4 cycles
- Arm B: Induction: Daunorubicin, cytarabine and midostaurin. Depending on response, second cycle of Induction may be given.
  Consolidation: High-dose cytarabine and midostaurin.
  Midostaurin: Induction: 50 mg orally twice daily x 14 days beginning on day 8
  Consolidation: 50 mg orally twice daily x 14 days beginning on day 8 of each cycle (up to 4 cycles)
  Daunorubicin: First Induction: Daunorubicin 90 mg/m²/day IV Days 1,2,3
  Second Induction, if needed: Daunorubicin 45 mg/m²/day IV Days 1,2,3
  Cytarabine: Induction: Cytarabine 100 mg/m²/day continuous infusion x 7 days starting Day 1
  Second Induction, if needed: Cytarabine 100 mg/m²/day continuous infusion x 7 days starting Day 1
  Consolidation: Cytarabine 3 g/m² (recommend 1.5 g/m² for age ≥ 55 or patients with decreased creatinine clearance) every 12 hours IV Days 1,3,5 or Days 1-3 for 6 doses for up to 4 cycles
Period: Overall Study
Arm/Group | Arm A | Arm B
Started | 90 | 87
Completed | 10 | 6
Not Completed | 80 | 81
Not completed — Adverse Event | 5 | 2
Not completed — Death | 4 | 1
Not completed — Lack of Efficacy | 7 | 10
Not completed — Physician Decision | 7 | 11
Not completed — Protocol Violation | 0 | 3
Not completed — Withdrawal by Subject | 2 | 10
Not completed — Intercurrent illness, Recurrence of disease, Subject proceeded to transplant or non-protocol therapy | 55 | 44

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 90 | 87 | 177
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (13) | 51 (12) | 51 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 54 | 103
  Male | 41 | 33 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 6 | 15
  Not Hispanic or Latino | 75 | 77 | 152
  Unknown or Not Reported | 6 | 4 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 7 | 8 | 15
  White | 69 | 68 | 137
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 11 | 8 | 19
ECOG (Eastern Cooperative Oncology Group) Performance Score [Count of Participants; unit: Participants] — 0: Fully active, able to carry on all pre-disease performance without restriction.
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature e.g. light house work, office work.
  2. Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours
  3. Capable of only limited self-care, confined to bed or chair more than 50% of waking hours
  4. Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair
  Participants
    0 | 22 | 22 | 44
    1 | 58 | 56 | 114
    2 | 8 | 7 | 15
    3 | 2 | 1 | 3
    Unknown | 0 | 1 | 1
AML Category [Count of Participants; unit: Participants] — De Novo AML: AML that develops spontaneously without prior blood disorders or cancer treatments. Often associated with a comparatively better prognosis
  Therapy-Related AML (t-AML): AML that arises as a result of previous chemotherapy or radiation therapy. Generally considered a higher-risk category
  AML with Myelodysplasia-Related Changes (AML-MRC): AML that originates from or shows features of prior myelodysplastic syndromes or dysplasia. Also associated with a worse prognosis compared to De Novo AML
  Participants
    AML with Myelodysplasia-Related Changes | 7 | 4 | 11
    De Novo AML | 80 | 79 | 159
    Therapy-Related AML | 3 | 4 | 7
WHO Classification [Count of Participants; unit: Participants]
  AML related to previous chemotherapy or radiation | 1 | 1 | 2
  AML with certain genetic abnormalities | 34 | 34 | 68
  AML with myelodysplasia-related changes | 5 | 2 | 7
  AML not otherwise specified | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: FLT3 Mutation Negative Composite Complete Response (CRc) [Includes Complete Response (CR) or CR With Incomplete Hematologic Recovery (CRi)] at End of Induction
Description: FLT3 mutation negative (evaluated by polymerase chain reaction [PCR]) Composite Complete Response (CRc) [includes CR and CRi] rate after induction treatment and complete MRD assessment. The cut points used for FLT3 mutation negative are 1% (equivalent to 10-2) for FLT3-TKD and 10-4 for FLT3-ITD.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 90 | 87
Participants | 36 | 41
Statistical Analysis 1: Comparison: Arm A vs Arm B; Test type: Superiority; p = 0.366, Fisher Exact — The threshold for statistical significance was p = 0.10; Proportion Difference = -0.071, 90% CI 2-sided [-0.205 to 0.062] — Treatment Difference = Arm A - Arm B

2. Secondary Outcome: FLT3 Mutation Negative Complete Response (CR) Rate at End of Induction
Description: CR evaluated by FLT3 testing after Induction
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 90 | 87
Participants | 33 | 37
Statistical Analysis 1: Comparison: Arm A vs Arm B; Test type: Superiority; p = 0.446, Fisher Exact — The threshold for statistical significance was p = 0.10; Proportion Difference = -0.059, 90% CI 2-sided [-0.191 to 0.073] — Treatment Difference = Arm A - Arm B

3. Secondary Outcome: Minimal Residual Disease (MRD)- CRc Rate at End of Induction
Description: MRD- CRc evaluated by flow cytometry after Induction
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 90 | 87
Participants | 58 | 52
Statistical Analysis 1: Comparison: Arm A vs Arm B; Test type: Superiority; p = 0.539, Fisher Exact — The threshold for statistical significance was p = 0.10; Proportion Difference = 0.047, 90% CI 2-sided [-0.084 to 0.178] — Treatment Difference = Arm A - Arm B

4. Secondary Outcome: CRc (CR or CRi) Rate at End of Induction
Description: CRc assessed in accordance with 2017 European LeukemiaNet (ELN)
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 90 | 87
Participants | 77 | 63
Statistical Analysis 1: Comparison: Arm A vs Arm B; Test type: Superiority; p = 0.042, Fisher Exact — The threshold for statistical significance was p = 0.10; Proportion Difference = 0.131, 90% CI 2-sided [0.020 to 0.242] — Treatment Difference = Arm A - Arm B

5. Secondary Outcome: Event Free Survival (EFS)
Description: EFS assessed in accordance with 2017 ELN
Time Frame: 68 months
Reporting Status: Not Posted

6. Secondary Outcome: Overall Survival (OS)
Description: OS assessed in accordance with 2017 ELN
Time Frame: 68 months
Reporting Status: Not Posted

7. Secondary Outcome: Number of Participants Treatment-related Adverse Events as Assessed by CTCAE v5.0
Description: Number of participants with abnormal laboratory values and/or adverse events
Time Frame: 10 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 90 | 87
Participants | 82 | 73

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) are monitored during the 9 month treatment period for each patient, and for 30 days post-final dose, until resolution to ≤ grade 1 or stabilization, for a total of 10 months.
Description: A serious adverse event (SAE) is any untoward medical occurrence after study treatment initiation that results in death, is life-threatening, requires or prolongs hospitalization, causes disability/incapacity, is a congenital anomaly, or, based on medical judgment, may jeopardize the patient or require intervention to prevent serious outcomes.
Arm/Group | Arm A | Arm B
All-Cause Mortality (participants affected / at risk) | 23/90 | 27/87
Serious Adverse Events (participants affected / at risk) | 48/90 | 39/87
Other Adverse Events (participants affected / at risk) | 83/90 | 81/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=90) | Arm B (N=87)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 2 (2) | 1 (1)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 1 (2) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 2 (2) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Neutropenic colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 4 (4)
Pneumonia (Infections and infestations) | 1 (2) | 2 (2)
Pneumonia fungal (Infections and infestations) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Sepsis (Infections and infestations) | 10 (10) | 2 (3)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis fungal (Infections and infestations) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Stomatitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Streptococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombophlebitis septic (Infections and infestations) | 1 (1) | 0 (0)
Troponin I increased (Investigations) | 0 (0) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1)
Cranial nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1)
Embolism venous (Vascular disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 2 (4) | 1 (1)
Escherichia sepsis (Infections and infestations) | 0 (0) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 24 (32) | 18 (23)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hypotension (Nervous system disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Oesophageal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Superficial vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=90) | Arm B (N=87)
Alanine aminotransferase increased (Investigations) | 16 (28) | 18 (36)
Anaemia (Blood and lymphatic system disorders) | 28 (158) | 34 (168)
Aspartate aminotransferase increased (Investigations) | 17 (24) | 24 (28)
Colitis (Gastrointestinal disorders) | 7 (8) | 5 (5)
Constipation (Gastrointestinal disorders) | 22 (23) | 9 (13)
Decreased appetite (Metabolism and nutrition disorders) | 15 (22) | 12 (13)
Diarrhoea (Gastrointestinal disorders) | 36 (44) | 25 (34)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 15 (19) | 8 (9)
Fatigue (General disorders) | 18 (23) | 17 (20)
Febrile neutropenia (Blood and lymphatic system disorders) | 48 (65) | 43 (58)
Hypocalcaemia (Metabolism and nutrition disorders) | 16 (29) | 7 (11)
Hypokalaemia (Metabolism and nutrition disorders) | 18 (33) | 28 (61)
Lymphocyte count decreased (Investigations) | 24 (179) | 26 (262)
Nausea (Gastrointestinal disorders) | 20 (27) | 22 (34)
Neutrophil count decreased (Investigations) | 28 (92) | 34 (151)
Platelet count decreased (Investigations) | 38 (292) | 33 (267)
Pyrexia (General disorders) | 16 (32) | 15 (31)
Sepsis (Infections and infestations) | 5 (5) | 9 (9)
Stomatitis (Gastrointestinal disorders) | 29 (33) | 25 (34)
Vomiting (Gastrointestinal disorders) | 11 (13) | 9 (11)
White blood cell count decreased (Investigations) | 31 (155) | 37 (225)
Abdominal pain (Gastrointestinal disorders) | 12 (14) | 11 (11)
Anxiety (Psychiatric disorders) | 7 (7) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0)
Bacteraemia (Infections and infestations) | 8 (10) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 6 (7) | 7 (15)
Blood bilirubin increased (Investigations) | 5 (6) | 6 (8)
Chills (General disorders) | 9 (9) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 0 (0)
Dizziness (Nervous system disorders) | 12 (12) | 6 (9)
Dry mouth (Gastrointestinal disorders) | 6 (6) | 0 (0)
Dysgeusia (Nervous system disorders) | 6 (6) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (12) | 6 (10)
Electrocardiogram QT prolonged (Investigations) | 6 (8) | 0 (0)
Flatulence (Gastrointestinal disorders) | 5 (5) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 6 (6)
Haematuria (Renal and urinary disorders) | 0 (0) | 6 (6)
Headache (Nervous system disorders) | 12 (15) | 10 (14)
Hyperphosphataemia (Metabolism and nutrition disorders) | 5 (6) | 0 (0)
Hypertension (Vascular disorders) | 9 (14) | 8 (10)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 8 (17) | 7 (16)
Hypomagnesaemia (Metabolism and nutrition disorders) | 9 (15) | 10 (24)
Hyponatraemia (Metabolism and nutrition disorders) | 7 (13) | 5 (6)
Hypophosphataemia (Metabolism and nutrition disorders) | 10 (17) | 17 (22)
Hypotension (Vascular disorders) | 11 (14) | 6 (8)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 7 (8)
Insomnia (Psychiatric disorders) | 10 (10) | 6 (6)
International normalised ratio increased (Investigations) | 0 (0) | 5 (9)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 5 (34)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 5 (16)
Neutropenia (Blood and lymphatic system disorders) | 6 (20) | 5 (25)
Oedema peripheral (General disorders) | 7 (10) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0)
Pneumonia (Infections and infestations) | 6 (6) | 5 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (7) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 7 (9) | 5 (6)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (9) | 8 (10)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 5 (5)
Syncope (Nervous system disorders) | 5 (7) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (46) | 7 (53)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-10-05): https://cdn.clinicaltrials.gov/large-docs/09/NCT03836209/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-09): https://cdn.clinicaltrials.gov/large-docs/09/NCT03836209/SAP_001.pdf